CLINICAL TRIAL: NCT04900909
Title: Health Status of Patients After Surgically Implanted Biological and Mechanical Aortic Valves: a Population-based Retrospective Analysis (2010-2018)
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Landesklinikum Sankt Polten (Other); Sicknessfund Burgenland (BGKK) (Unknown); A.ö. Krankenhaus St. Josef Braunau GmbH (Other)
Responsible Party: Principal Investigator, Hendrik Jan Ankersmit, Principal Investigator/Univ. Prof. , MD, MBA, Medical University of Vienna
Other Study IDs: AUTHEARTVISIT
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Aortic valve replacement with mechanical valves
  Interventions: Device: Aortic Valve Replacement
- Aortic valve replacement with bioprostheses
  Interventions: Device: Aortic Valve Replacement

INTERVENTIONS:
Device: Aortic Valve Replacement — Surgical replacement of aortic valves

SUMMARY:
The overall project aim is to study outcomes following aortic valve replacement with either mechanical valves or bioprostheses by retrieving data from the main social security carriers in Austria for the years 2010-2018.

DETAILED DESCRIPTION:
The purpose of this research project is to evaluate mortality (primary outcome) and incidence of heart attack, stroke, reoperation and first diagnosis of heart insufficiency (secondary outcomes) after aortic valve replacement. We aim to compare those outcomes between mechanical valves and bioprostheses.

Data will be retrieved from the main social security carriers in Austria (covering 98% of its population) from 2010-2018.

ELIGIBILITY:
Inclusion Criteria:

* isolated surgical aortic valve replacement in Austria

Exclusion Criteria:

* below 18 years of age
* concomitant heart surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent isolated surgical aortic valve replacement in Austria above 18 years of age with no other concomitant heart surgery were included.
Sampling Method: Non-Probability Sample
Enrollment: 13993 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 8 years
  all cause mortality after aortic valve replacement

SECONDARY OUTCOMES:
reoperation | 8 years
  incidence of reoperation after aortic valve replacement
stroke | 8 years
  incidence of stroke after aortic valve replacement
heart attack | 8 years
  incidence of heart attack after aortic valve replacement
heart insufficiency | 8 years
  incidence of heart insufficiency after aortic valve replacement

IPD SHARING:
Plan to Share IPD: No